CLINICAL TRIAL: NCT04187183
Title: Use of Fresh Platelet-rich Plasma With Concentrated Leukocytes or Fresh Platelet-rich Plasma Without Concentrated Leukocytes for Treating Knee Cartilage Degeneration: a Randomized Controlled Trial
Brief Title: Use of Fresh Platelet Rich Plasma With Concentrated Leukocytes or Fresh Platelet Rich Plasma Without Concentrated Leukocytes in the Treatment of Knee Cartilage Degeneration: a Randomized Controlled Trial
Acronym: PRP019
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRP019
Record Dates: First submitted 2019-11-27; First posted 2019-12-05 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Leukocyte Count

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fresh PRP with concentrate Leukocyte (Experimental): Three infiltrations of fresh Platelet Rich Plasma with concentrated Leukocytes
  1 infiltration weekly, for 3 weeks.
  Interventions: Other: Fresh Platelet Rich Plasma with leukocyte
- Fresh PRP without concentrated Leukocyte (Active Comparator): Three infiltrations of fresh Platelet Rich Plasma without concentrated Leukocyte.
  1 infiltration weekly, for 3 weeks.
  Interventions: Other: Fresh Platelet Rich Plasma without leukocyte

INTERVENTIONS:
Other: Fresh Platelet Rich Plasma with leukocyte — autologous Platelet Rich Plasma with leukocyte will be infiltrate in the knee joint
  Arms: Fresh PRP with concentrate Leukocyte
Other: Fresh Platelet Rich Plasma without leukocyte — autologous Platelet Rich Plasma without leukocyte will be infiltrate in the knee joint
  Arms: Fresh PRP without concentrated Leukocyte

SUMMARY:
The aim of the study is to compare the triple infiltration of Fresh Platelet Rich Plasma with concentrated Leukocytes against triple infiltration of Fresh Platelet Rich Plasma Without Concentrated Leukocytes in the treatment of Knee Cartilage Degeneration in a Double Blind Randomized Controlled Trial

DETAILED DESCRIPTION:
Platelet Rich Plasma has a consolidated use in the field of orthopedic surgery to reduce inflammation, promoting bone regeneration and healing of surgical wounds.

Some clinical studies demonstrated the utility of the intra-articular infiltration of Platelet Rich Plasma in the treatment of knee articular cartilage lesions, becoming a common conservative strategies in the management of these diseases.

Actually, there are some different kinds of PRP formulations, in particular, the scientific debate is focusing on the role of Leukocytes and if it is better using fresh or frozen PRP.

At the moment don't exist randomized controlled clinical studies comparing fresh PRP rich in Leukocyte against PRP poor in Leukocyte in the treatment of knee cartilage lesions.

The study has two groups of patients, the first will undergo to three infiltrations of Fresh Platelet Rich Plasma With Concentrated Leukocytes and the second will undergo to three infiltrations of Fresh Platelet Rich Plasma Without Concentrated Leukocytes, each infiltrations will be done weekly.

ELIGIBILITY:
Inclusion Criteria:

Patients with degenerative pathology of the knee cartilage with:

1. Age between 18 and 75 years;
2. Unilateral involvement;
3. Signs and symptoms of degenerative pathology of the cartilage of the knee;
4. Radiographic or MRI signs of degenerative pathology of the cartilage of the knee (Kellgren-Lawrence 1-4 degrees);
5. Hemoglobin> 11 g / dl; Platelet count> 150,000 plt / mm3 (recently performed blood count);
6. No clinically significant electrocardiographic alteration (recently performed ECG).
7. Patients' ability and consent to actively participate in clinical follow-up;
8. Signature of informed consent.

Exclusion Criteria:

1. Patients undergone to intra-articular infiltration of another substance in the previous 6 months;
2. Patients undergone knee surgery in the previous 12 months;
3. Patients with malignant neoplasms;
4. Patients suffering from rheumatic diseases;
5. Patients suffering from diabetes;
6. Patients with hematologic diseases (coagulopathies);
7. Patients on anti-anticoagulant therapy;
8. Patients suffering from thyroid metabolic disorders;
9. Patients abusing alcoholic beverages, drugs or drugs;
10. Body Mass Index> 35;
11. Patients who have taken NSAIDs within 3 days before taking blood;
12. Patients with cardiovascular diseases for which the 150 ml blood test would be contraindicated;
13. Patients with a recently performed blood count with Hb values <11 g / dl and Platelets <150,000 plt / mm3.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2024-10-03 (Actual); Study Completion 2024-10-03 (Actual)

PRIMARY OUTCOMES:
IKDC-subjective score (International Knee Documentation Committee) | 12 month
  It is a specific subjective rating scale for te knee. Iti s one of the most reliable tools for assessing knee diseases. The survey examines three categories: symptoms, sport activity, knee function.

SECONDARY OUTCOMES:
KOOS score (Knee Injury and Osteoarthritis Outcome Score) | baseline, 2, 6, 12 and 24 months
  KOOS consists of 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL). The previous week is the time period considered when answering the questions. Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale
EQ-VAS (EuroQol-visual analogue scales) | baseline, 2, 6, 12, 24 months
  It is a rating scale for assessing the health state of the patient. The scale ranging from 0 (the worst health state) to 100 (the best health state)
EQ-5D (EuroQoL) Current Health Assessment | baseline, 2, 6, 12, 24 months
  It is a reliable tools for assessing quality of life of the patient
Tegner Activity Level Scale | baseline, 2, 6, 12, 24 months
  Survey useful for assessing sport activity of the patient. The Tegner activity scale is a one-item score that graded activity based on work and sports activities on a scale of 0 to 10. Zero represents disability because of knee problems and 10 represents national or international level soccer.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

REFERENCES:
- [Background] Di Martino A, Di Matteo B, Papio T, Tentoni F, Selleri F, Cenacchi A, Kon E, Filardo G. Platelet-Rich Plasma Versus Hyaluronic Acid Injections for the Treatment of Knee Osteoarthritis: Results at 5 Years of a Double-Blind, Randomized Controlled Trial. Am J Sports Med. 2019 Feb;47(2):347-354. doi: 10.1177/0363546518814532. Epub 2018 Dec 13. PMID 30545242
- [Background] Everts PA, Knape JT, Weibrich G, Schonberger JP, Hoffmann J, Overdevest EP, Box HA, van Zundert A. Platelet-rich plasma and platelet gel: a review. J Extra Corpor Technol. 2006 Jun;38(2):174-87. PMID 16921694
- [Background] Sanchez AR, Sheridan PJ, Kupp LI. Is platelet-rich plasma the perfect enhancement factor? A current review. Int J Oral Maxillofac Implants. 2003 Jan-Feb;18(1):93-103. PMID 12608674
- [Background] Filardo G, Kon E, Pereira Ruiz MT, Vaccaro F, Guitaldi R, Di Martino A, Cenacchi A, Fornasari PM, Marcacci M. Platelet-rich plasma intra-articular injections for cartilage degeneration and osteoarthritis: single- versus double-spinning approach. Knee Surg Sports Traumatol Arthrosc. 2012 Oct;20(10):2082-91. doi: 10.1007/s00167-011-1837-x. Epub 2011 Dec 28. PMID 22203046
- [Background] Cavallo C, Filardo G, Mariani E, Kon E, Marcacci M, Pereira Ruiz MT, Facchini A, Grigolo B. Comparison of platelet-rich plasma formulations for cartilage healing: an in vitro study. J Bone Joint Surg Am. 2014 Mar 5;96(5):423-9. doi: 10.2106/JBJS.M.00726. PMID 24599205
- [Background] Assirelli E, Filardo G, Mariani E, Kon E, Roffi A, Vaccaro F, Marcacci M, Facchini A, Pulsatelli L. Effect of two different preparations of platelet-rich plasma on synoviocytes. Knee Surg Sports Traumatol Arthrosc. 2015 Sep;23(9):2690-703. doi: 10.1007/s00167-014-3113-3. Epub 2014 Jun 19. PMID 24942296
- [Derived] Romandini I, Boffa A, Di Martino A, Andriolo L, Cenacchi A, Sangiorgi E, Orazi S, Pizzuti V, Zaffagnini S, Filardo G. Leukocytes Do Not Influence the Safety and Efficacy of Platelet-Rich Plasma Injections for the Treatment of Knee Osteoarthritis: A Double-Blind Randomized Controlled Trial. Am J Sports Med. 2024 Nov;52(13):3212-3222. doi: 10.1177/03635465241283500. Epub 2024 Oct 12. PMID 39394763